CLINICAL TRIAL: NCT06856473
Title: Effects of Dry Needling on Spasticity and Functional Ability in Children With Cerebral Palsy
Brief Title: Effects of Dry Needling on Spasticity and Functional Ability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Responsible Party: Principal Investigator, Mohamed A. Abdel Ghafar, Professor, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMCDryNeedle
Record Dates: First submitted 2025-02-23; First posted 2025-03-04 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy (CP)
Keywords: Dry Needle; Spasticity; Functional abilities
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: The study follows a randomized controlled trial (RCT) design with a parallel-group interventional model to evaluate the effects of dry needling on spasticity and functional outcomes. Participants are randomly assigned to one of two groups:
  Study Group (Intervention Group): Receives dry needling for the spastic calf and adductor muscles in addition to a traditional physical therapy program based on Neurodevelopmental Treatment (NDT) (3 sessions per week, each lasting 1 hour).
  Control Group: Receives only the traditional physical therapy program (NDT) without dry needling, following the same frequency and duration.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional physical therapy Group (Active Comparator): Traditional physical therapy program based on neurodevelopmental treatment (NDT) (3 sessions per week, each lasting 1 hour).
  Interventions: Other: Traditional Physical Therapy
- Dry needling Group (Experimental): traditional physical therapy program based on neurodevelopmental Treatment (NDT) (3 sessions per week, each lasting 1 hour), in addition to dry needling for the spastic calf and adductor muscles.
  Interventions: Other: Traditional Physical Therapy; Other: Dry Needling

INTERVENTIONS:
Other: Traditional Physical Therapy — Traditional Physical Therapy based on neurodevelopmental technique
  Other Names: Conventional physical therapy
Other: Dry Needling — Dry Needling in addition to the same traditional physical therapy program
  Other Names: Study group
  Arms: Dry needling Group

SUMMARY:
This study investigates the effects of dry needling on spasticity and its impact on functional ability in individuals with neuromuscular disorders. Using the Modified Ashworth Scale (MAS), Timed Up and Go (TUG) test, and Gross Motor Function Measure (GMFM), the research evaluates changes in muscle tone, mobility, and overall motor performance following dry needling intervention. The findings aim to provide evidence on the clinical benefits of dry needling as a therapeutic approach for improving movement efficiency and functional outcomes in patients with spasticity.

DETAILED DESCRIPTION:
Spasticity is a common impairment in individuals with neuromuscular disorders, often leading to limitations in movement, balance, and overall functional performance. Dry needling has emerged as a promising intervention for managing spasticity by targeting hyperactive muscle fibers and reducing abnormal muscle tone. This study aims to explore the therapeutic effects of dry needling on muscle spasticity and functional ability using standardized clinical measures.

Participants will undergo pre- and post-intervention assessments using the Modified Ashworth Scale (MAS) to quantify changes in muscle tone, the Timed Up and Go (TUG) test to evaluate mobility and balance, and the Gross Motor Function Measure (GMFM) to assess functional motor skills. The intervention will focus on specific muscle groups affected by spasticity.

By analyzing the relationship between changes in spasticity and functional mobility, this study seeks to determine whether dry needling contributes to measurable improvements in movement efficiency, postural control, and daily functional activities. The findings will provide valuable insights into the role of dry needling as an adjunct therapy in rehabilitation programs, supporting its integration into clinical practice for individuals with neuromuscular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Hypertonia score 2 according to MAS
* Able to understand and follow instructions
* Able to stand and walk independantly

Exclusion Criteria:

* Participants with neurological conditions that involve significant cognitive deficits or severe uncontrolled epilepsy
* Participants who have undergone surgical procedures within the last 3 months

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Modified Ashwarth Scale (MAS) | Week 12 after intervention completion
  The MAS measures spasticity on a 6-point ordinal scale from 0 to 4, with an additional 1+ category. Minimum Value (0): No increase in muscle tone (better outcome). Maximum Value (4): Affected part(s) rigid in flexion or extension (worse outcome). Higher scores indicate greater spasticity, representing a worse outcome.

SECONDARY OUTCOMES:
Gross Motor Function Measure (GMFM) | Week 12 after intervention completion.
  The GMFM is scored on a 0 to 100% scale, reflecting the percentage of motor tasks successfully performed. Minimum Value (0%): No motor function achieved (worse outcome). Maximum Value (100%): Full achievement of all motor tasks (better outcome). Higher scores indicate better gross motor function and improved mobility.
Time up and go test (TUG) | Week 12 after intervention completion
  The TUG test measures the time (in seconds) taken to stand up from a chair, walk 3 meters, turn around, walk back, and sit down. Minimum Value (lower time in seconds): Faster completion time indicates better mobility and functional performance. Maximum Value (higher time in seconds): Slower completion time indicates impaired mobility and a higher risk of falls (worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- BMC, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No